CLINICAL TRIAL: NCT01834781
Title: Transcranial Pulsed Electromagnetic Fields for Multiple Chemical Sensitivity: a Study Protocol for a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Pulsed Electromagnetic Fields for Multiple Chemical Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Danish Research Centre for Chemical Sensitivities (Other)
Collaborators: Aage Bangs Fond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCS-Re5
Record Dates: First submitted 2013-04-12; First posted 2013-04-18 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Chemical Sensitivity
Keywords: multiple chemical sensitivity, re5 therapy, pulsed electromagnetic fields
MeSH Terms: conditions — Multiple Chemical Sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulsed electromagnetic fields (Active Comparator): Pulsed electromagnetic fields is applied transcranially 30 minutes twice a day for 7 days a week over 6 consecutive weeks
  Interventions: Device: Pulsed electromagnetic fields
- Wearing the inactive device (Placebo Comparator): The inactive device is worn on the head for 30 minutes twice a day for 7 days a week over 6 consecutive weeks
  Interventions: Device: w/o pulsed electromagnetic fields

INTERVENTIONS:
Device: Pulsed electromagnetic fields
  Other Names: Re5 Independent System; Re5 therapy
  Arms: Pulsed electromagnetic fields
Device: w/o pulsed electromagnetic fields
  Arms: Wearing the inactive device

SUMMARY:
The purpose of this study is to determine whether pulsed electromagnetic fields(PEMF) is effective in the treatment of multiple chemical sensitivity in terms of life impact, symptoms, psychological distress, markers of central sensitization and the immune system, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Lacour's criteria for multiple chemical sensitivity
* Lifestyle or functional impairments that score ≥ 35 on the Life Impact scale of the Quick Environmental Exposure and Sensitivity Inventory
* Signed informed consent

Exclusion Criteria:

* previous PEMF therapy
* psychosis or a comparable disorder
* epilepsy
* cerebral tumours
* leukaemia or malignancies in the head or neck region
* having a pacemaker or other active implants
* pregnancy or nursing
* unreliable contraception
* drug or alcohol abuse
* a pending application or intentions to apply for early retirement
* initiation of pharmacological treatment which have not steadied
* participation in another research study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Life Impact Scale (Quick Environmental Exposure and Sensitivity Inventory) | Week 1, 2, 3, 4, 5, 6, and 2½ and 4½ month follow-ups
  The Life Impact Scale is part of the Quick Environmental Exposure and Sensitivity Inventory (QEESI). The QEESI consists of five scales measuring different domains related to chemical sensitivities, i.e. commonly reported symptoms, chemical (inhalant) intolerances, other intolerances, life impact attributed to chemical intolerances, and on-going exposures from routinely used products (Masking Index). The Life Impact Scale consists of 10 items, where responses are rated on an 11 point scale ranging from "not at all a problem" (0) to "disabling symptoms" (10)), resulting in a score range from 0 to 100.

SECONDARY OUTCOMES:
Change from baseline in Symptom Severity Scale (Quick Environmental Exposure and Sensitivity Inventory) | Week 1, 2, 3, 4, 5, 6, and 2½ and 4½ month follow-ups
  The Symptom severity scale from the QEESI consist of ten items where responses are rated on an eleven point scale ranging from "not at all a problem" (0) to "disabling symptoms" (10), resulting in a score range from 0 to 100.
Change from baseline in Chemical Intolerance Scale (Quick Environmental Exposure and Sensitivity Inventory) | Week 1, 2, 3, 4, 5, 6, and 2½ and 4½ month follow-ups
  The Chemical Intolerance scale from the QEESI consist of ten items where responses are rated on an eleven point scale ranging from "not at all a problem" (0) to "disabling symptoms" (10), resulting in a score range from 0 to 100.
Change from baseline in Sheehan Disability Scale | Week 1, 2, 3, 4, 5, 6, and 2½ and 4½ month follow-ups
  The Sheehan Disability Scale (SDS) is widely used in psychiatry, but has also been applied to many other chronic medical illnesses. It uses visuo-spatial, numeric and descriptive anchors to measure impaired functioning in three domains: work, social life and family life. The scale generates four disability scores, one for each domain and a total score by adding up the three individual domain scores
Change from baseline in individual self-selected tasks | Week 1, 2, 3, 4, 5, 6, and 2½ and 4½ month follow-ups
  In addition to the Life Impact scale used as the primary outcome measure, the participants will need to select three tasks in the areas of work, social life and family life, which are impaired by MCS at baseline. The degree of impairment associated with each task is scored on a scale from 0-10 with visuo-spatial, numeric and descriptive anchors similar to SDS.
Change from baseline in noise sensitivity | Week 6, and 2½ and 4½ month follow-ups
  To measure the participants' sensitivity to noise, they will be asked to grade their responses to 10 different noises (e.g. drone of a machine, stroke of a hammer, rustling of paper) on a 5-point Likert scale.
Change from baseline in depression (Symptom Check List-92) | Week 1, 2, 3, 4, 5, 6, and 2½ and 4½ month follow-ups
  The Symptom Checklist 92 (SCL-92) subscales for depression, anxiety and somatization will be included. These subscales comprise 35 items on which responses are rated on a 5-point Likert scale ranging from not at all to very much.
Change from baseline in anxiety (Symptom Check List-92) | Week 1, 2, 3, 4, 5, 6, and 2½ and 4½ month follow-ups
Change from baseline in somatization (Symptom Check List-92) | Week 1, 2, 3, 4, 5, 6, and 2½ and 4½ month follow-ups
Change from baseline in 6-item Hamiltons Depression Scale | Week 1, 2, 3, 4, 5, 6, and 2½ and 4½ month follow-ups
  The 6-item Hamilton Depression Rating Scale (HAM-D6) is a short self-administered measure of depression. The scale has been shown to be as sensitive as the more widely used 17-item Hamilton Depression Rating Scale (HAM-D17) to measure antidepressive treatment effects.
Change from baseline in Perceived Stress Scale | Week 1, 2, 3, 4, 5, 6, and 2½ and 4½ month follow-ups
  The short version of the Perceived Stress Scale (PSS-10) consists of 10 questions and measures the self-perception of stress by grading how different life situations are perceived. The PSS-10 has been shown to be a valid and reliable measure of perceived stress.
Change from baseline in World Health Organization Quality Of Life Brief version | Week 6 and 4½ month follow-ups
  The brief version of World Health Organization Quality Of Life (WHOQOL-BREF) is a short multidimensional questionnaire, which measures health-related quality of life. The scale consists of four domains: physical health, psychological well-being, social relationships and environment.
Change from baseline in capsaicin-induced secondary punctate hyperalgesia | Week 6
Change from baseline in immunological markers in serum | Week 6
  IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, IL-17, IL-21, IL-22, IL-23, TNFα, IFNγ

CONTACTS AND LOCATIONS:
Locations (1):
- The Danish Research Centre for Chemical Sensitivities, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Tran MT, Skovbjerg S, Arendt-Nielsen L, Christensen KB, Elberling J. Transcranial pulsed electromagnetic fields for multiple chemical sensitivity: study protocol for a randomized, double-blind, placebo-controlled trial. Trials. 2013 Aug 16;14:256. doi: 10.1186/1745-6215-14-256. PMID 23947742